CLINICAL TRIAL: NCT00082199
Title: A Randomized, Multicenter, Double-Blind, Placebo Controlled Study of the Efficacy and Safety of Aripiprazole in the Maintenance of Abstinence From Alcohol in Subjects With Alcoholism
Brief Title: Study of Aripiprazole in Subjects With Alcoholism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka America Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CN138-089
Record Dates: First submitted 2004-04-30; First posted 2004-05-04 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2008-07

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Aripiprazole

ARMS (2):
- A1 (Active Comparator)
  Interventions: Drug: Aripiprazole
- A2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aripiprazole — Tablets, Oral, 2-30mg, Once daily, 12 weeks.
  Other Names: Abilify
  Arms: A1
Drug: Placebo — Tablets, Oral, Once daily, 12 weeks.
  Arms: A2

SUMMARY:
The purpose of this clinical research study is to learn whether subjects treated with aripiprazole are able to abstain from alcohol use for a greater number of days than subjects treated with placebo. The safety of using aripiprazole will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of alcohol dependence who want to stop using alcohol will be considered for the study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2004-04; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Assessment of abstinence from the consumption of alcohol during the study

SECONDARY OUTCOMES:
Assessment of alcohol use during the study and behavioral measures of substance abuse an dependence

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (14):
- United States (14):
  - Local Institution, Farmington, Connecticut
  - Local Institution, New Haven, Connecticut
  - Local Institution, Indianapolis, Indiana
  - Local Institution, Boston, Massachusetts
  - Local Institution, New York, New York
  - Local Institution, Rochester, New York
  - Local Institution, Chapel Hill, North Carolina
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Providence, Rhode Island
  - Local Institution, Charleston, South Carolina
  - Local Institution, Dallas, Texas
  - Local Institution, Houston, Texas
  - Local Institution, Charlottesville, Virginia
  - Local Institution, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Anton RF, Kranzler H, Breder C, Marcus RN, Carson WH, Han J. A randomized, multicenter, double-blind, placebo-controlled study of the efficacy and safety of aripiprazole for the treatment of alcohol dependence. J Clin Psychopharmacol. 2008 Feb;28(1):5-12. doi: 10.1097/jcp.0b013e3181602fd4. PMID 18204334